CLINICAL TRIAL: NCT06743282
Title: Senyo Health App - Connecting Primary Care to Substance Use Disorder Treatment Using a Telehealth Collaborative Care Platform
Brief Title: Senyo Health With Substance Use Disorder (SUD) in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tyler S. Oesterle, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-007758; 1R18HS029774-01 (AHRQ)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senyo (Experimental): Subjects to the Senyo group will begin receiving intervention immediately, and will move to the follow-up phase after 12 weeks.
  Interventions: Behavioral: Senyo App; Behavioral: Follow-up

INTERVENTIONS:
Behavioral: Senyo App — Subjects will engage with the Senyo Health platform for 12 weeks to deliver Integrated Behavioral Healthcare (IBH) treatment. The Senyo Health platform consists of asynchronous cognitive behavioral therapy modules and weekly check-ins with the IBH care manager. Subjects will also complete a monthly urine test for substances, the Timeline Follow Back (TLFB) to gather substance abuse history, and complete weekly questionnaires.
Behavioral: Follow-up — Subjects will have monthly check-in meetings with the Integrated Behavioral Healthcare manager, complete monthly urine tests for substance use, the Timeline Follow Back (TLFB) to gather substance abuse history, and complete monthly questionnaires.

SUMMARY:
The purpose of this study is to examine the barriers, facilitators, and optimal processes for implementing a digitally enhanced screening, brief intervention, and referral to treatment (SBIRT) model for Substance Use Disorder SUD treatment among Mayo primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, write, and understand English
* Minimum DAST (1+), audit-C score (3+)
* Access and willingness to use a mobile device for asynchronous (text) and synchronous (video) engagement with care.
* Access to or willingness to obtain a Primary care provider at a participating Mayo Clinic site;
* Eligibility determined by ASAM Assessment

Exclusion Criteria:

* Diagnosed personality pathology as the primary presenting concern based on clinical judgment, severe cognitive impairment (e.g., intellectual disability or dementia), or psychosis
* Inability to actively participate in and learn from psychotherapeutic interaction based on clinical evaluation and clinical judgment
* Needing a higher level of mental health care as demonstrated by ASAM32 assessment.
* Decline to answer suicidality questions.
* Already admitted into or about to initiate treatment in another addiction treatment program.

Currently attending High School.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Substance Craving Scale (BSCS) | Baseline, weekly for 12 weeks, 4 months, 5 months, 6 months
  The Brief Substance Craving Scale is a 16 item, self-report instrument that assesses craving for substances of abuse over a 24 hour period. Intensity and frequency of craving are recorded on a five-point Likert scale, with 0 = Not at all, 1 = Slight, 2 = Moderate, 3 = Considerable, and 4 = Extreme.
Timeline Follow Back | Baseline, weekly for 12 weeks, 4 months, 5 months, 6 months
  Timeline Follow Back is an assessment to document substance use over a specific period of time

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, weekly for 12 weeks, 4 months, 5 months, 6 months
  The General Anxiety Disorder 7-item (GAD 7) scale to assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, weekly for 12 weeks, 4 months, 5 months, 6 months
  The Patient Health Questionnaire 9-item (PHQ-9) scale used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Oesterle, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oesterle TS, Bormann NL, Paul MM, Breitinger SA, Lai B, Smith JL, Stoppel CJ, Arndt S, Williams MD. Treatment of Substance Use Disorders With a Mobile Phone App Within Rural Collaborative Care Management (Senyo Health): Protocol for a Mixed Methods Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 26;14:e65693. doi: 10.2196/65693. PMID 40138685